CLINICAL TRIAL: NCT00001058
Title: A Phase II/III Prospective, Multicenter, Randomized, Controlled Trial Comparing the Safety and Efficacy of Three Clarithromycin-Containing Combination Drug Regimens for the Treatment of Disseminated Mycobacterium Avium Complex (MAC) Disease in Persons With AIDS
Brief Title: A Comparison of Three Drug Combinations Containing Clarithromycin in the Treatment of Mycobacterium Avium Complex (MAC) Disease in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 223; 11200 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Clofazimine; Acquired Immunodeficiency Syndrome; Ciprofloxacin; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Indinavir; Ritonavir; Ethambutol; Clarithromycin; Rifabutin

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Rifabutin

SUMMARY:
To compare the efficacy and safety of clarithromycin combined with rifabutin, ethambutol, or both in the treatment of disseminated Mycobacterium avium Complex (MAC) disease in persons with AIDS, including individuals who have or have not received prior MAC prophylaxis.

It is believed that effective therapy for MAC disease in patients with AIDS requires combinations of two or more antimycobacterial agents in order to overcome drug resistance and the unfavorable influence of the profound immunosuppression associated with AIDS. Data suggest that clarithromycin may have substantial activity in two- or three-drug combination regimens with clofazimine, rifamycin derivatives, ethambutol, or the 4-quinolones.

DETAILED DESCRIPTION:
It is believed that effective therapy for MAC disease in patients with AIDS requires combinations of two or more antimycobacterial agents in order to overcome drug resistance and the unfavorable influence of the profound immunosuppression associated with AIDS. Data suggest that clarithromycin may have substantial activity in two- or three-drug combination regimens with clofazimine, rifamycin derivatives, ethambutol, or the 4-quinolones.

Patients are randomized to one of three treatment arms containing clarithromycin in combination with ethambutol, rifabutin, or both. Clarithromycin alone is taken on days 1 through 3 to determine tolerance and rifabutin and/or ethambutol is added on day 3. AS PER AMENDMENT 7/2/97: Patients may elect to add ritonavir or indinavir to their treatment regimen. Treatment continues daily for 48 weeks. In the absence of a dose-limiting toxicity, those patients who are determined to be complete or partial responders continue on the regimen to which they were originally assigned. Patients who have failed or relapsed on originally assigned MAC therapy, must have their therapy amended to receive clarithromycin and at least two other drugs not included in their originally assigned regimen. Patients are followed twice in the first week, then every 2 weeks for the first 2 months, then monthly for the next 4 months, and then every 2 months thereafter until the end of 12 months. PER AMENDMENT 10/10/96: NOTE: Any patient who develops a toxicity to rifabutin or ethambutol after week 12 or thereafter will be offered the option of being registered to a salvage regimen of 2 new drugs not previously received, plus clarithromycin to continue for the study duration.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Maintenance or prophylactic therapy for other opportunistic infections (with the exception of specifically excluded drugs).
* Carbamazepine or theophylline.
* Isoniazid for TB prophylaxis.

PER AMENDMENT 10/10/96:

* Therapy for acute infectious processes, other than MAC, provided that the patient is stable on the therapy.
* Fluconazole therapy for maintenance or suppression of fungal infections, providing the patient has been on a stable dose for at least 4 weeks.

PER AMENDMENT 7/02/97:

* If a patient elects to receive indinavir, ORTHO/NOVUM 1/35 is an acceptable means of birth control.

Patients must have:

* HIV infection.
* Disseminated MAC disease.
* Life expectancy of at least 8 weeks.
* Consent of parent or guardian if under 18 years of age.

NOTE:

* This protocol is approved for prisoner participation.

Prior Medication:

Allowed:

PER AMENDMENT 10/10/96:

* Therapy for acute infectious processes, other than MAC, prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active mycobacterial infection other than MAC that requires treatment, with the exception of isoniazid used solely for TB prophylaxis.

Concurrent Medication:

Excluded:

* Other antimycobacterial drugs (with the exception of isoniazid for TB prophylaxis).
* Other investigational drugs unless approved by protocol chair.

PER AMENDMENT 7/2/97:

* For patients who elect to receive indinavir or ritonavir:
* Terfenadine, astemizole, cisapride, triazolam, or midazolam.
* For patients who elect to receive ritonavir:
* alprazolam, amiodarone, bepridil, bupropion, cisapride, clorazepate, clozapine, diazepam, dihydroergotamine, ergotamine, estazolam, encainide, flecainide, flurazepam, meperidine, pimozide, piroxicam, propafenone, propoxyphene, quinidine or zolpidem.
* For patients who elect to receive indinavir:
* oral contraceptives other than ORTHO/NOVUM as a sole form of birth control.
* For patients randomized to a rifabutin-containing arm:
* oral contraceptives or Norplant as a sole form of birth control.

Patients with the following prior condition are excluded:

* History of severe hypersensitivity to erythromycin, clarithromycin, azithromycin, ethambutol, rifampin, or rifabutin (including Type 1 hypersensitivity reaction, Stevens-Johnson syndrome, hepatitis, optic neuritis, or exfoliative dermatitis).

Prior Medication:

Excluded:

* Empiric or presumptive antimycobacterial therapy prior to study entry if > 14 days, within 90 days prior to entry.

NOTE:

* Patients unwilling to discontinue presumptive therapy or empiric therapy may be enrolled with the permission of the protocol chairs, however, if they are without a MAC positive blood culture at baseline, they will have study medications discontinued (AS PER AMENDMENT 7/2/97).

PER AMENDMENT 10/10/96:

* Treatment with clarithromycin or ethambutol within 4 days of initiation of study medications.
* Treatment with rifabutin or rifampin within 7 days of initiation of study medications.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246
Dates: Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benson CA, Study Chair; Chaisson RE, Study Chair; Currier JS, Study Chair
Locations (34):
- United States (33):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Flexner C, Noe D, Benson C, Currier J, Andrade A, Shaver A. Adherence patterns in patients with symptomatic Mycobacterium avium complex (MAC) infection taking a twice-daily clarithromycin regimen. ACTG 223 Study Team. Int Conf AIDS. 1998;12:585 (abstract no 32324)
- [Background] Benson CA, Williams PL, Currier JS, Holland F, Mahon LF, MacGregor RR, Inderlied CB, Flexner C, Neidig J, Chaisson R, Notario GF, Hafner R; AIDS Clinical Trials Group 223 Protocol Team. A prospective, randomized trial examining the efficacy and safety of clarithromycin in combination with ethambutol, rifabutin, or both for the treatment of disseminated Mycobacterium avium complex disease in persons with acquired immunodeficiency syndrome. Clin Infect Dis. 2003 Nov 1;37(9):1234-43. doi: 10.1086/378807. Epub 2003 Oct 3. PMID 14557969